CLINICAL TRIAL: NCT06613802
Title: Prevalence of Gabapentinoids in Geriatric Falls Outpatients in Aalborg in 2013-2014, 2018-2019, and 2023
Brief Title: Prevalence of Gabapentinoids and Opioids in Geriatric Falls Patients
Status: Completed | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Johannes Riis, Professor, Aalborg University Hospital
Other Study IDs: F2024-085
Record Dates: First submitted 2024-09-12; First posted 2024-09-26 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-01

CONDITIONS: Gabapentin
MeSH Terms: interventions — Time

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- 2013-2014: Patients in 2013-2014. All fall patient charts will be included depending on the prevalence of gabapentionoid prescriptions. It is expected that the prevalence in 2013 is twice (6%) that of the background population (3%). Sample size calculations at 80% power and 5% significance based on differences in population between 2023 (estimated 20%, which is twice that of 2023 background population of 10%) shows that 90 participants are required. Thus it is expected to include the whole of 2013. However, if the prevalence is lower than expected, 2014 will also be included. The sample size required prevalences of 3% in 2013 and 10% in 2023 is 194, which would be met by expanding the sampling frame to encompass 2014.
  Interventions: Other: Time
- 2018-2019: All patients in 2018 will be included. If it is necessary to also include 2014 as described above, then 2019 will also be included to ensure approximately equal group sizes.
  Interventions: Other: Time
- 2023: More patients were seen in 2023, with a total of 254 available. If only 2013 is included based on the prevalence as stated above, then every second patient from 2023 will be included. If 2014 is also included then all patient from 2023 will be included to ensure approximately equal group sizes.
  Interventions: Other: Time

INTERVENTIONS:
Other: Time — This is a cross sectional study, and the exposure where the outcome is expected to change by is time. Years included in the study are 2013-2014, 2018-2019 and 2023

SUMMARY:
This study investigates the prescription patterns of gabapentinoids (gabapentin and pregabalin) in a geriatric fall clinic in Aalborg, Denmark, between 2013 and 2023. Gabapentinoids, often prescribed for neuropathic pain, have seen increased off-label usage, particularly as alternatives to opioids. Despite the lack of robust evidence supporting their efficacy in many neuropathic and non-neuropathic pain conditions, their use has grown, especially in elderly populations. This raises concerns about their potential side effects, such as drowsiness, dizziness, and the risk of falls, especially when combined with opioids.

The study aims to determine the prevalence of gabapentinoid and opioid prescriptions in the clinics and for what type of pain they are prescribed. Furthermore, the study will look into the development in opioid prescriptions and concomitant gabapentinoid/opioid usage in this population.

The study is a retrospective chart review of patient charts from the years 2013-2014, 2018-2019, and 2023, analyzing patient characteristics, comorbidities, medication lists, and pain classifications.

ELIGIBILITY:
Inclusion Criteria:

* patient in the geriatric fall clinic at Aalborg University Hospital in either 2013-2014, 2018-2019, or 2023

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The entire sample will be included. It is expected that the prevalence in 2013 is twice (6%) that of the background population (3%). Sample size calculations at 80% power and 5% significance based on differences in population between 2023 (estimated 20%, which is twice that of 2023 background population of 10%) shows that 90 participants are required. Thus it is expected to include the whole of 2013, 2018 and every second patient in 2023 based on this. However, if the prevalence is lower than expected in 2013 then 2014, 2019 and all patients in 2023 will be included.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of gabapentionoids | Baseline. That is at the time of first outpatient contact in the geriatric fall clinic at Aalborg University Hospital
  Number of patients taking gabapentinoids (yes/no) for each year
Prevalence of opioids | Baseline. That is at the time of first outpatient contact in the geriatric fall clinic at Aalborg University Hospital
  Number of patients taking opioids (yes/no) for each year

SECONDARY OUTCOMES:
Pain characteristics for each year | Baseline. That is at the time of first outpatient contact in the geriatric fall clinic at Aalborg University Hospital
  Pain categorized as malignant, neuropathic (with subcategories such as radiculopathy, postherpetic neuralgia), nociceptive somatic (e.g., back pain, shoulder pain), and nociceptive visceral (e.g., headache, abdominal pain). Each pain type will further be classified by duration as acute (below 3 months), subacute (3-6 months), chronic (more than 6 months), or "not stated in charts".

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided